CLINICAL TRIAL: NCT01420536
Title: A Cross-over Randomized Clinical Trial of Canine Guidance and Bilateral Balanced Occlusion in Complete Denture Wearers
Brief Title: Canine Guidance vs Bilateral Balanced Occlusion in Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Raphael Freitas de Souza, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Unesp-PT-001; 2008/07183-5 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2011-08-10; First posted 2011-08-19 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: Bilateral Balanced Occlusion; Canine Guidance; Complete Denture; Denture Retention; Dental Occlusion; Edentulous; Edentulism; Mandibular movement; Mastication; Patient Acceptance of Health Care; Patient Satisfaction
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous; Bites and Stings; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canine Guidance (Experimental): Complete dentures adjusted with "mutually protected articulation in which the vertical and horizontal overlap of the canine teeth disengage the posterior teeth in the excursive movements of the mandible" (The Glossary of Prosthodontic Terms. J. Prosthet. Dent., 94(1): 10-92)
  Interventions: Procedure: Occlusal scheme
- Bilateral Balanced Occlusion (Sham Comparator): Complete dentures as conventionally adjusted: anterior and posterior teeth presented bilateral contact in excentric positions
  Interventions: Procedure: Occlusal scheme

INTERVENTIONS:
Procedure: Occlusal scheme — Before enrollment, all participants will receive conventional complete dentures adjusted according to the bilateral balanced occlusion concept.
  Following randomization, canine guidance will be achieved by adding composite resin (Restorative Z100, 3M Brazil, Sumaré, SP, Brazil) on the lingual surface of the maxillary canines. A sham comparator will also employ the addition of composite, but without changing eccentric contacts.
  Other Names: Dental articulation; Denture oclusion

SUMMARY:
The objective of this study is to compare the canine guidance (CG) and bilateral balanced occlusion (BBO) on denture satisfaction and kinesiographic parameters of complete denture wearers, by means of a cross-over trial. Edentulous patients will receive new maxillary and mandibular complete dentures and, after the intraoral adjustments and adaptation period, will randomly receive a sequence of occlusal schemes: BBO followed by CG, or CG followed by BBO.

DETAILED DESCRIPTION:
Reference for published version of the complete study:

Paleari AG, Marra J, Rodriguez LS, De Souza RF, Pero AC, De A Mollo Jr F, Compagnoni MA. A cross-over randomised clinical trial of eccentric occlusion in complete dentures.J Oral Rehabil. 2012 Apr 9. doi: 10.1111/j.1365-2842.2012.02299.x. [Epub ahead of print]

ELIGIBILITY:
Inclusion Criteria:

* Adult patients needing new complete dentures
* Mentally receptiveness
* Absence of dysfunctional disorders of the masticatory system
* Normal volume and resilience of residual edentulous ridges
* Absence of debilitating systemic diseases

Exclusion Criteria:

* Use of cardiac pacemaker
* Refusal to participate or inability to provide informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael F de Souza, DDS, PhD, Principal Investigator — University of Sao Paulo; Marco A Compagnoni, DDS, PhD, Study Director — Araraquara Dental School -Universidade Estadual Paulista (Sao Paulo State University)
Locations (1):
- Araraquara Dental School -Universidade Estadual Paulista (Sao Paulo State University), Araraquara, São Paulo, Brazil

REFERENCES:
- [Derived] Paleari AG, Marra J, Rodriguez LS, de Souza RF, Pero AC, Mollo Fde A Jr, Compagnoni MA. A cross-over randomised clinical trial of eccentric occlusion in complete dentures. J Oral Rehabil. 2012 Aug;39(8):615-22. doi: 10.1111/j.1365-2842.2012.02299.x. Epub 2012 Apr 9. PMID 22486470
- See also: Institutional page of the Araraquara Dental School (research site) — http://www.foar.unesp.br
- See also: Institutional page of the Ribeirão Preto Dental School (PI's institution ) — http://www.forp.usp.br
- See also: Principal Investigator´s CV (RF Souza) — http://lattes.cnpq.br/7092555880664311
- See also: Study director´s CV (MA Compagnoni) — http://lattes.cnpq.br/8921196002764597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July to December 2012. Convenience sample composed by 50 patients, who had volunteered to receive new complete dentures at Araraquara Dental School - UNESP.
Pre-assignment Details: Participants waited 30 days following the completion of treatment, in order to have them functionally adapted to their new dentures. Six spontaneously declined to participate before random assignment due to lack of interest.
Groups:
- Canine Guidance, Then Bilateral Balanced Occlusion: Canine guidance: Complete dentures adjusted with "mutually protected articulation in which the vertical and horizontal overlap of the canine teeth disengage the posterior teeth in the excursive movements of the mandible" (The Glossary of Prosthodontic Terms. J. Prosthet. Dent., 94(1): 10-92); Bilateral Balanced Occlusion: Complete dentures as conventionally adjusted, i.e. anterior and posterior teeth presented bilateral contact in excentric positions
- Bilateral Balanced Occlusion, Then Canine Guidance: Bilateral Balanced Occlusion: Complete dentures as conventionally adjusted, i.e. anterior and posterior teeth presented bilateral contact in excentric positions; Canine guidance: Complete dentures adjusted with "mutually protected articulation in which the vertical and horizontal overlap of the canine teeth disengage the posterior teeth in the excursive movements of the mandible" (The Glossary of Prosthodontic Terms. J. Prosthet. Dent., 94(1): 10-92).
Period: Period 1 (30 Days)
Arm/Group | Canine Guidance, Then Bilateral Balanced Occlusion | Bilateral Balanced Occlusion, Then Canine Guidance
Started | 22 | 22
Completed | 19 (Participants declined to participate further before changing interventions.) | 22
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0
Period: Period 2 (30 Days)
Arm/Group | Canine Guidance, Then Bilateral Balanced Occlusion | Bilateral Balanced Occlusion, Then Canine Guidance
Started | 19 | 22
Completed | 19 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bilateral Balanced Occlusion Then Canine Guidance: Bilateral Balanced Occlusion: Complete dentures as conventionally adjusted, i.e. anterior and posterior teeth presented bilateral contact in excentric positions; Canine guidance: Complete dentures adjusted with "mutually protected articulation in which the vertical and horizontal overlap of the canine teeth disengage the posterior teeth in the excursive movements of the mandible" (The Glossary of Prosthodontic Terms. J. Prosthet. Dent., 94(1): 10-92);
- Total: Total of all reporting groups
Arm/Group | Canine Guidance, Then Bilateral Balanced Occlusion | Bilateral Balanced Occlusion Then Canine Guidance | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.6) | 66.4 (10.3) | 66.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Brazil | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Denture Satisfaction
Description: Assessed by a questionnaire questionnaire based on the criteria used by Celebic and Knezovic-Zlataric (A comparison of patient's satisfaction between complete and partial removable denture wearers. J Dent. 2003;21:445-451) and used by Souza et al. (Validation of the Brazilian versions of two inventories for measuring oral health-related quality of life of edentulous subjects. Gerodontology. 2012;29:e88-95.).
  Eight questions were answered according to a three-point scale (0=unsatisfactory; 1=regular; 2=good), whose sum provided a summary satisfaction score that ranged from 0 (the participant is completely dissatisfied with existing dentures) to 16 (maximum satisfaction).
Time Frame: 30 days
Population: Convenience sampling.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Canine Guidance: Canine guidance: Complete dentures adjusted with "mutually protected articulation in which the vertical and horizontal overlap of the canine teeth disengage the posterior teeth in the excursive movements of the mandible" (The Glossary of Prosthodontic Terms. J. Prosthet. Dent., 94(1): 10-92)
- Bilateral Balanced Occlusion: Bilateral Balanced Occlusion: Complete dentures as conventionally adjusted, i.e. anterior and posterior teeth presented bilateral contact in excentric positions
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
units on a scale | 15 [12 to 16] | 15 [12 to 16]
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; Statistical analysis was performed by a researcher who was unaware of all procedures performed. The questionnaire about denture satisfaction originated a general score that was compared using the Wilcoxon test, according to the two tested conditions; Test type: Superiority or Other; p = 0.569, Wilcoxon (Mann-Whitney) — P values less than 0.05 would be considered statistically significant in this study

2. Secondary Outcome: Kinesiographic Parameters -- (1.a) Maximum Mouth Opening, Vertical Axis
Description: Mandibular physiologic movements and the pattern of maxillary denture movement during chewing, as recorded by a kinesiograph (K6-I Diagnostic System, Myotronics research Inc., Seatle, WA).
  Specific measures involved: (1) Mouth opening; (2) Movement of the mandible from rest position to maximal occlusion (tooth clenching position); (3) Movement of the mandible during chewing; and (4) Movement of the upper denture base during chewing. Data from each measure was not combined into new variables, and collected in a single time point after each intervention.
  All measures were taken according to the vertical, anteroposterior and left-right axes separately.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 30.3 (4.5) | 30.9 (4.6)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; For the kinesiographic assessment, the Kolmogorov-Smirnov test was used to evaluate whether the variables had normal distribution, which was positive in the majority of cases. A comparison between the values obtained for both groups was performed by means of the paired sample t-test; Test type: Superiority or Other; p = 0.339, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

3. Secondary Outcome: Kinesiographic Parameters -- (1.b) Maximum Mouth Opening, Anteroposterior Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 25.1 (9.4) | 25.8 (8.8)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.515, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

4. Secondary Outcome: Kinesiographic Parameters -- (1.c) Maximum Mouth Opening, Left-right Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 1.4 (1.3) | 1.7 (2.4)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.485, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t test

5. Secondary Outcome: Kinesiographic Parameters -- (2.a) Rest Position, Vertical Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 2.1 (1.2) | 2.3 (1.1)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.111, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

6. Secondary Outcome: Kinesiographic Parameters -- (2.b) Rest Position, Anteroposterior Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 1.9 (1.0) | 1.9 (0.9)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.399, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

7. Secondary Outcome: Kinesiographic Parameters -- (2.c) Rest Position, Left-right Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 0.5 (0.5) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.550, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

8. Secondary Outcome: Kinesiographic Parameters -- (3.a) Mandibular Chewing Movement, Vertical Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 12.0 (2.7) | 12.1 (2.7)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.609, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

9. Secondary Outcome: Kinesiographic Parameters -- (3.b) Mandibular Chewing Movement, Anteroposterior Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 4.2 (2.1) | 4.3 (2.0)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.600, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

10. Secondary Outcome: Kinesiographic Parameters -- (3.c) Mandibular Chewing Movement, Left-right Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | 1.2 (2.1) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.611, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

11. Secondary Outcome: Kinesiographic Parameters -- (4.a) Upper Denture Base Movement, Vertical Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | -0.5 (0.4) | -0.6 (0.3)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.044, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

12. Secondary Outcome: Kinesiographic Parameters -- (4.b) Upper Denture Base Movement, Anteroposterior Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | -0.4 (0.7) | -0.4 (0.4)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.677, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

13. Secondary Outcome: Kinesiographic Parameters -- (4.c) Upper Denture Base Movement, Left-right Axis
Description: as for outcome 2
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Number analyzed (Participants) | 39 | 39
mm | -0.1 (0.5) | -0.1 (0.3)
Statistical Analysis 1: Comparison: Canine Guidance vs Bilateral Balanced Occlusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.885, t-test, 2 sided — P values less than 0.05 would be considered statistically significant in this study; Paired t-test

ADVERSE EVENTS:
Arm/Group | Canine Guidance | Bilateral Balanced Occlusion
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/44 | 0/41

LIMITATIONS AND CAVEATS:
* Losses during follow-up (although only 3 participants declined to continue the research - relatively small number);
* Possibility of errors in the kinesiographic assessment (low and equally distributed between the different conditions).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No